CLINICAL TRIAL: NCT02299531
Title: Effects of Portion Size and Energy Density of a Single Meal in Preschool Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Barbara J. Rolls, Professor of Nutrition and Director of The Laboratory for the Study of Human Ingestive Behavior, Penn State University
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: ChildFood201; R01DK082580 (NIH)
Record Dates: First submitted 2014-11-19; First posted 2014-11-24 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Feeding Behaviors
MeSH Terms: conditions — Feeding Behavior | interventions — Portion Size

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Low Energy Density, Small Portions (Experimental): Low meal energy density and small portion sizes
  Interventions: Other: Varying meal energy density and portion size
- Low Energy Density, Medium Portions (Experimental): Low meal energy density and medium portion sizes
  Interventions: Other: Varying meal energy density and portion size
- Low Energy Density, Large Portions (Experimental): Low meal energy density and large portion sizes
  Interventions: Other: Varying meal energy density and portion size
- High Energy Density, Small Portions (Experimental): High meal energy density and small portion sizes
  Interventions: Other: Varying meal energy density and portion size
- High Energy Density, Medium Portions (Experimental): High meal energy density and medium portion sizes
  Interventions: Other: Varying meal energy density and portion size
- High Energy Density, Large Portions (Experimental): High meal energy density and large portion sizes
  Interventions: Other: Varying meal energy density and portion size

INTERVENTIONS:
Other: Varying meal energy density and portion size

SUMMARY:
This study investigates the effect of varying both energy density and portion size of all foods at lunch on preschool children's intake. The foods used in this study are commercially-available, commonly-consumed foods with typical variations in energy density. The primary aim of the study is to investigate the independent and combined effects of energy density and portion size on preschool children's intake at a meal composed of foods typically served to this population.

ELIGIBILITY:
Inclusion Criteria:

* Children must be enrolled in participating childcare centers.

Exclusion Criteria:

* Allergy or intolerance to any of the foods or beverages served.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 131 (Actual)
Dates: Start 2013-05; Primary Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Food and energy intake (Food weight (grams) and energy (kcal) | Once a week for four weeks

SECONDARY OUTCOMES:
Meal energy density (Energy density (kcal/g) | Once a week for four weeks
  Energy density (kcal/g)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J Rolls, PhD, Principal Investigator — Penn State University
Locations (1):
- The Pennsylvania State University, Laboratory for the Study of Human Ingestive Behavior, University Park, Pennsylvania, United States

REFERENCES:
- [Derived] Kling SM, Roe LS, Keller KL, Rolls BJ. Double trouble: Portion size and energy density combine to increase preschool children's lunch intake. Physiol Behav. 2016 Aug 1;162:18-26. doi: 10.1016/j.physbeh.2016.02.019. Epub 2016 Feb 12. PMID 26879105